CLINICAL TRIAL: NCT04569591
Title: Desmopressin (DDAVP) Stimulation for 18F-FDG-PET Detection of Pituitary Adenoma in Cushing's Disease
Brief Title: Corticotrophin-releasing Hormone (CRH) Stimulation for 18F-FDG-PET Detection of Pituitary Adenoma in Cushing s Disease
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 200048; 20-N-0048
Record Dates: First submitted 2020-09-29; First posted 2020-09-30 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2025-11-21

CONDITIONS: Cushing's Disease; Pituitary Adenoma
Keywords: Corticotropinoma; Pituitary Microadenoma; Acthrel
MeSH Terms: conditions — Pituitary ACTH Hypersecretion; Pituitary Neoplasms | interventions — corticorelin ovine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 1 (Experimental): patients aged 8 or older with Cushing's Disease who are surgical candidates for resection of ACTH producing pituitary adenoma within 12 weeks of PET imaging
  Interventions: Drug: Acthrel

INTERVENTIONS:
Drug: Acthrel — Intravenous administration of ovine CRH (Acthrel (Registered Trademark) 1 mcg/kg up to a maximum dose of 100 mcg) results in selective increase in ACTH activity of pituitary adenomas within two minutes and peaks between 10-15 minutes.

SUMMARY:
Background:

Cushing s disease is caused by a pituitary gland tumor. Patients with Cushing s disease suffer obesity, diabetes, osteoporosis, weakness, and hypertension. The cure is surgery to remove the pituitary tumor. Currently, MRI is the best way to find these tumors. But not all tumors can be seen with an MRI. Researchers hope giving the hormone CRH before a PET scan can help make these tumors more visible.

Objective:

To test whether giving CRH before a PET scan will help find pituitary gland tumors that might be causing Cushing s disease.

Eligibility:

People ages 8 and older with Cushing s disease that is caused by a pituitary gland tumor that cannot be reliably seen on MRI

Design:

Participants will be screened with their medical history, a physical exam, an MRI, and blood tests.

Participants will have at least one hospital visit. During their time in the hospital, they will have a physical exam and a neurological exam. They will have a PET scan of the brain. A thin plastic tube will be inserted into an arm vein. A small amount of radioactive sugar and CRH will be injected through the tube. Participants will lie in a darkened room for about an hour and be asked to urinate. Then they will lie inside the scanner for about 40 minutes. After the scan, they will be asked to urinate every 2-3 hours for the rest of the day. Blood will be drawn through a needle in the arm.

Participants will have surgery to remove their tumor within 3 months after the scan.

Participants will then continue regular follow-up in the clinic.

DETAILED DESCRIPTION:
Study Description:

This study is designed as a single institution trial. The study utilizes safe and clinically-validated tools for preoperative workup of subjects with small pituitary tumors. DDAVP stimulation and 18F-labeled fluorodeoxyglucose (FDG) uptake for PET-imaging will be used to detect MRInegative pituitary adenomas in subjects with Cushing s disease. Subjects who have MRI-negative pituitary microadenomas will undergo FDG PETimaging with DDAVP stimulation. Intravenous FDG will be given approximately four hours following DDAVP administration. Within 24 weeks after completion of the FDG high-resolution PET scan, subjects will undergo surgical resection of the pituitary adenoma. Surgical and histological confirmation of adenoma location will be noted. All images will be read independently by neuroradiologists blinded to clinical and histopathological outcomes. The diagnostic and localization accuracy of PET-imaging will be assessed by comparing the PET findings with histopathology.

Objectives:

Cushing s disease (CD) affects 3,000 people in the United States every year and results in significant morbidity and early mortality. The disease is caused by millimeter sized pituitary microadenomas (corticotropinomas) that secrete adrenocorticotropic hormone (ACTH). Surgical resection of corticotropinomas remains the most effective treatment strategy. Preoperative magnetic resonance imaging (MRI) can detect microadenomas in approximately 50-80% of subjects. Subjects with microadenomas invisible on MR imaging are exposed to more invasive explorations of the sella with fewer instances of hormone remission and higher complications. Corticotropinomas can be detected by FDG positron emission tomography (PET) in 50% of subjects. Prior work by us suggests that secretagogue stimulation with corticotropin-releasing hormone (CRH) leads to increased FDG uptake and improved PET detection of pituitary microadenomas.

Since, CRH is no longer available, we will use DDAVP which has a similar biological activity to CRH. If validated, DDAVP-stimulated FDG-PET imaging could provide a complementary imaging modality to improve visualization of ACTH-secreting microadenomas and surgical planning.

Primary Objective:

The primary objective of this study is to determine the detection rate of MRI-negative pituitary adenomas in subjects with Cushing's disease by DDAVP-stimulated FDG PET imaging. We will analyze whether or not DDAVP-stimulated PET imaging demonstrates

tumor in MRI-negative cases by assessing the accuracy and sensitivity of high-resolution FDG PET-imaging detection of ACTH-adenomas that could not be reliably detected on MR-imaging.

Secondary Objectives:

To assess the accuracy of FDG high-resolution PETimaging localization of ACTH-adenomas in CD compared to surgical and

histologic localization. This will be achieved by comparing actual tumor location confirmed by histological findings during surgical resection to the location predicted by PET- and MR-imaging within subjects.

Endpoints:

Primary Endpoint: The primary outcome measure will be defined as whether or not DDAVP-stimulated PET imaging demonstrates tumor in MRI-negative cases. This will be demonstrated by assessing the accuracy and sensitivity of FDG high-resolution PET-imaging detection of ACTH-adenomas that could not be reliably detected on MR-imaging.

Secondary Endpoints: Location of tumor on preoperative PET-imaging and location of tumor during surgery. Histopathological confirmation of ACTH-adenoma will be the gold-standard to measure the primary and secondary endpoints.

ELIGIBILITY:
* INCLUSION CRITERIA:

In order to be eligible to participate in this study, an individual must meet all of the following criteria:

1. Subjects aged 8 or older with biochemical evidence of Cushing s disease and a clinical MRI pituitary neuroradiology result of negative or possible adenoma (e.g. "no tumor" or "possible tumor")
2. MRI of the pituitary gland with and without contrast obtained within 9 months of screening
3. For newly diagnosed Cushing s disease cases, IPSS is required.
4. Ability to undergo PET-imaging without general anesthesia
5. Ability to provide informed consent for study participation (parents or guardians in the case of minors)
6. Clinical diagnosis of Cushing s disease based on documented medical records
7. Surgical candidate for and subject agrees to resection of ACTH producing pituitary adenoma within 24 weeks of PET-imaging
8. Normal liver function as evidenced by liver enzyme tests completed within 14 days before injection of radiopharmaceutical: SGOT, SGPT <= 5 x upper limit of normal; bilirubin <= 2 x upper limit of normal

EXCLUSION CRITERIA:

An individual who meets any of the following criteria will be excluded from participation in this study:

1. Pregnancy or lactation
2. Glomerular filtration rate < 50 mL/min/1.73 m^2, hepatorenal syndrome, history of urinary retention or post-liver or kidney transplantation.
3. Hyponatremia (serum sodium below 135 mmol/L)
4. A history of angina, significant coronary artery disease, congestive heart failure, or SIADH due to risk of fluid overload and/or hyponatremia.
5. Uncontrolled hypertension (blood pressure >150/95 mmHg) due to risk of further increase if fluid overload occurs.
6. Uncontrolled, severe hypotension (sustained blood pressure <90/60), or symptomatic hypotension.
7. Current use of any of the following medications:

   * Vasopressors: phenylephrine, dopamine and vasopressin.
   * Drugs that can worsen hyponatremia:

   non-steroidal anti-inflammatory drugs (NSAIDs) within 4 days of testing, loop diuretics (bumetanide, ethacrynic acid, furosemide, torsemide), chlorpromazine, chlorpropamide, cisplatin, monoamine oxidase inhibitors (MAOI), opiate agonists, oxybutynin, selective serotonin reuptake inhibitors (SSRI), vincristine, tricyclic antidepressants (TCA),

   -Drugs that interfere with DDAVP duration of action or potency:

   carbamazepine, lamotrigine, tolvaptan
8. Habitual or psychogenic polydipsia, due to increased risk of hyponatremia
9. History of Type IIB von Willebrand s disease due to risk for thrombosis.
10. Elevated blood glucose level above 200 mg/dL on the day of the scan prior to FDG administration.
11. Known intolerance to DDAVP

INCLUSION OF VULNERABLE PARTICIPANTS:

* Children: Children age 8 and older are included in this protocol. More than half of the subjects with CD requiring transsphenoidal surgery at the NIH are children. The knowledge gained by the use of DDAVP PET imaging in children with MR-invisible tumors will provide generalizable knowledge in the treatment of CD in this population. Children under the age of 8 usually require anesthesia for a PET scan, which involves greater risk. Therefore, children under the age of 8 will be excluded from participation.
* Pregnant or lactating women: Pregnant and lactating women will be excluded from participation. The PET radiopharmaceutical used in this study can be harmful to a developing fetus. Therefore women who are able to become pregnant will have a pregnancy test performed within 24 hours before PET imaging. Individuals will not be able to participate in PET scanning if the pregnancy test results positive.

Ages: 8 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2026-02-09 (Estimated); Primary Completion 2026-04-20 (Estimated); Study Completion 2026-04-20 (Estimated)

PRIMARY OUTCOMES:
CRH-stimulated PET imaging demonstrates tumor in MRI-negative cases. | Baseline
  The primary outcome measure will be defined as whether or not CRH- stimulated PET imaging demonstrates tumor in MRI-negative cases. This will be demonstrated by assessing the accuracy and sensitivity of 18F-FDG high-resolution PET-imaging detection of ACTH-adenomas that could not be reliably detected on MR-imaging. Measures will include determining the rate of true tumor detection using PET-imaging compared to histologically-confirmed tumor location.

SECONDARY OUTCOMES:
Elevation of SUV of 18F-FDG | Baseline
  To measure the elevation of SUV of 18F-FDG within adenomas compared to surrounding normal gland following CRH stimulated PET imaging.

CONTACTS AND LOCATIONS:
Overall Officials: Prashant Chittiboina, M.D., Principal Investigator — National Institute of Neurological Disorders and Stroke (NINDS)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2020-N-0048.html